CLINICAL TRIAL: NCT06188091
Title: Impact of Active Joint Movement to Increase Range of Motion in Knee Joint After Primary or Revision Total Knee Arthroplasty
Brief Title: Joint Movement to Increase Range of Motion in Knee Joint After Primary Total Knee Arthroplasty
Acronym: ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22020545
Record Dates: First submitted 2023-12-05; First posted 2024-01-03 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-09

CONDITIONS: Total Knee Arthroplasty
Keywords: Range of motion; Physical therapy; Rehabilitation; Patient monitored exercises; Active mobilization exercises; Movement exercises; Mobility training; Mobility exercises; Flexion exercises; Stretching; Extension exercises; Movement therapy; Improved range of motion; ROM; Improved function; Active range of motion; Knee function; Active Range of movement
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All patients admitted to the hospital because of a knee problem are assign to a date of hospitalizing in random order by the secretary.
  Once at the hospital the knee patients, who might be candidates for the enrollment of the study, will get the ROM of the knees measured by a blinded physiotherapist trained in measuring knee joint.
  After joint measuring, there will be held a drawing from a bag which contains equal numbers marked either with a 2 or 8. The number is only known by the principal investigator and the 2 therapist who will introduce the patients to the exercises and instruct in the daily interval of doing the exercises (2 or 8). The therapist invites the patients which meets the inclusion criteria to take part in the study.
  After 18 days of treatment the outcome assessors will once again measure the ROM on patients included in the study (same therapist that did the the first measuring of a specific patient)
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor: Have no knowledge of the intervention the individual patient has received Participant, are asked to join after they meet the criteria's for inclusion, they know what intervention they get but no knowledge of the intervention in the other group Care Provider - know at the time for the first intervention right after drawing number 2 or 8
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention with active exercises for knee joint 2 times a day (Active Comparator): Intervention group A does 1 active exercise to improve flexion and 1 active exercise to improve extension 2 times a day, 18 days in a row
  Interventions: Behavioral: Exercise
- Intervention with active exercises for knee joint 8 times a day (Active Comparator): Intervention group B does 1 active exercise to improve flexion and 1 active exercise to improve extension 8 times a day, 18 days in a row
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Physiotherapeutic instructions to patients to do active exercise to improve the mobility of knee joint post-surgical

SUMMARY:
The goal of this clinical trail is to investigate if specific active exercises, with a certain daily frequency improves the range of motion (ROM) in the knee joint after primary- or revision total knee arthroplasty (TKA)

The main questions it aims to answer are:

* Does it make a difference to the ROM of the knee joint to do specific active exercise 2 times a day compared to 8 times a day in an 18 days period of time
* Analyze if range of motion in the knee joint after TKA has an impact on self-reported activity, pain and physical activity

Participants will be instructed by a physiotherapist to do a specific exercise to improve the flexion of the knee-joint and and other to improve the extension of the knee-joint.

One group will be instructed to do the exercises 2 times a day the other group to do the exercises 8 times a day in total of 18 days

The two groups will be compared to see if there is an effect in ROM and if the effect is significant between the groups if the intervention is done 2 times versus 8 times a day.

DETAILED DESCRIPTION:
There is a lack of knowledge about specific rehabilitation in relation to improving joint mobility of the knee joint, especially in terms of frequency and the active roll of the patients. The studies available describe predominantly passive joint mobilization after TKA (machine/therapist). Therefore there is a lack of knowledge about specific training methods regarding how patients can actively help increase joint mobility.

The purpose of the study is to verify whether increased frequency of two specific active joint movement exercises, for reduced flexion and/or extension, respectively, at fixed daily intervals over a continuous 18-day period can further increase joint mobility after TKA.

The hypothesis is that patients can increase joint mobility after TKA by repeating individual movement exercises with a high daily frequency.

Based on previous clinical experience at the department and data from published articles, a realistic assessment is that patients who receive intervention with a high frequency of joint movement exercises (8 times daily) will be able to achieve an increased flexion of approx. 12 degrees compared to low-frequency intervention (2 times daily), where it is estimated that flexion can be increased by 4 degrees from baseline. Thus, there will be a change between the two intervention groups of 8 degrees.

If this kind of focused movement training has an effect, it will have a major impact on the composition of postoperative rehabilitation.

Montebello is a department for specialized rehabilitation under North Zealand Hospital, Capital Region of Denmark. Patients are referred by doctors after determining the need for specialized rehabilitation due to a complicated course of the disease. Thus, it is patients who are accessed as needing a more intensive and specialized course than a usual general rehabilitation offers under municipal communities.

Every year, approx. 1675 patients are received within various specialties, of which between 250-300 patients are referred for knee care.

Thus, knee patients who are referred for admission to Montebello have all experienced complications in relation to their knee function. This can be severe fractures, complicated joint/cartilage damage, TKA with reduced mobility and subsequent brisement, or revision TKA due to infection or anything else related to replacement of the osteosynthesis material.

Intervention Both groups participate in exercise program based on group training in groups of 11 patients focused on improving knee function. The general training consists of strength, conditioning, balance, coordination, walking and movement training. Exercises are adjusted according to the individual's physical level and pain intensity. The daily frequency of physical exercise is between 2-4 sessions per day (approx. 45 minutes per session).

In addition, instruction is given in appropriate training in relation to prosthesis and pain management, education in strength and stability training, instruction in the use of TENS (Transcutaneous Electric Nerve Stimulation).

Both groups will receive supervision/instruction from the therapist about specific joint movement exercises to be performed on their own.

Short-term and long- term risks:

During the exercise, patients may experience pain/tightening. It is normal for irritation of the knee joint to occur after the exercises. This irritation must have subsided before the next round of practice.

Should it turn out that the patient cannot complete 2 or 8 repetitions without increased pain intensity, they are excluded from the project. Experience from the clinic shows that very few patients cannot complete the exercises many times a day. Retrospectively, it is estimated that approx. 20 patients out of approx. 2000 have not been able to complete the exercises due to increased pain. It is very unlikely that the patients will have any long-term negative side effects from preforming the exercises.

Collection of data Both intervention and control groups have their active joint mobility (ROM) of the knee joint on day 1 for exercise as well as day 18 for hospitalization.

Measurement of ROM and secondary outcome is carried out by physiotherapists affiliated with other specialties in the department, and thus do not have knowledge of which intervention group the individual patient belongs to. Drawing for the intervention group takes place after data has been collected. Therapists who perform measurements and tests also do not participate in the daily training of patients.

Before the start of the examination, the therapist who performs joint measurements will be trained in the procedure for measuring according to the chosen method to ensure optimal reliability of the measurement. The same physiotherapist will be measuring the ROM at day 1 and day 18 on the specific patient.

Therapists who measure ROM and perform the other tests are instructed not to ask the patient what intervention they have received during the re-testing process. Likewise, the patient is instructed not to talk about the intervention himself.

The selected manual for measuring knee joint mobility by goniometer has been validated. A goniometer with a 30 cm arm shall be used.

It is assumed that a difference of more than 5°represents a real clinical change in the same test.

ROM is measured on the 1st day of training at 8.15 am and immediately afterwards other functional tests are performed. On the 18th day of training, measurements and tests are repeated at the same time.

All measurements and tests performed on patients are already well known to therapists and are used daily on the ward.

Statistics and analysis Baseline consists of measurements of ROM, as well as the other of the numeric outcome variables collected on the 1st day of training.

Measurements from the two intervention groups are compared against each other. Paired t-tests will be performed for each of the intervention groups. Unpaired t-test is used to test for change between the two intervention groups. Results are considered significant when p<0.05. Analysis of data will be carried out in the IBM SPSS Statistics.

Sample size is calculated based on the expectation of 8° degree difference between low intensity compared to high intensity of movement exercises (4° vs. 12°). Standard deviation taken from 2018 department data (data from patients with lack of flexion 105° or less). Number in the two intervention groups 1-1, Power 80% and significance level 5%.

In this way, it is calculated that in each intervention group there must be 30 patients and 20% (6 persons) to ensure size in case of dropout a total of 36. However, as a solid data basis is desired, the goal is to strengthen the study by including a total of 50 patients in each group.

Ethics and data security Patients participating in this trial do not receive treatment that exposes them to invasive procedures, new medication, or otherwise exposes them to greater risk than the treatment normally included in the rehabilitation of TKA patients on the ward. The intervention is exercises that are already included in many places in the rehabilitation of TKA patients and are generally used among physiotherapists as good clinical practice after TKA.

The patients are informed that they can withdraw his or her consent at any time.

Processing of personal data in the project:

The study has been approved by the Danish Data Protection Agency. The collected data will be stored according to rules of the data protection agency in the Capital Region. All project data collected, will be handled in accordance with the rules of the Capital Region, in relation to current legislation. No data are sent abroad.

Funding The initiative to plan and execute the study is done by physiotherapist and development- and quality coordinator on the ward. Support in terms of advice and statistical analyses are given from the research department at NOH. There are no funding outside of the NOH and additional time used to execute the study is covered within the ward.

No remuneration is paid to the project participants.

Presentation of results The result should have interest to physiotherapist and orthopedic medical staff interested in rehabilitation after total knee arthroplasty both in Denmark and internationally.

The study results will be presented in an article aim to be published in national and international peer reviewed journals and in public media. Both positive, negative and inconclusive results will be published. The study will be registered at www.clinicaltrails.

Internally, at the ward at NOH, the results will be used to evaluate and reflect on the practice of current rehabilitation. Depending of the results it might have influence on the rehabilitation offered to patients with primary-or revision total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria

* Primary or revision total knee arthroplasty
* 105° or less Flexion in knee joint;
* Last post operation date 6 weeks to 6 month

Exclusion Criteria

* Unilateral arthroplasty in knee joint
* Other operations in knee joint than total knee arthroplasty
* Flexion in knee joint more than 105°
* Operation more than 6 month ago

Randomizing: The visitation team assesses all referrals coming from doctors (orthopedic surgeons, general practitioners, private practice specialists) and accepts those patients for admission who are within the visitation guidelines. No members of the visitation have direct patient contact in relation to the training at Montebello. Patients are accepted through the Health Platform (SP) used in the Capital Region of Denmark.

After visitation, secretaries will summon patients to planned knee teams on available dates. The secretaries are geographically located 3000 kilometers away from the department and have no knowledge of the research project. In chronological order, in relation to the time of visitation, patients will be summoned to a given date. As there can be a maximum of 11 patients on a given admission date, others awaiting admission will be allocated the next available date and so on.

Due to the department's continuous reception of patients, where up to 11 knee patients are received in the same team on a given date, randomization cannot take place at a individual level but at team-level, so that patients hospitalized on the same date do not receive two different interventions since they train together during the 3 weeks.

When the actual admission takes place and the patient is physically at Montebello, a joint measurement of the knee joint will be performed by the therapist (this is not part of the project group and does not instruct knee patients). Based on this joint measurement and the other inclusion criteria, relevant patients for the project will be invited to take part in the study and included with consent.

Whether a group of patients receives intervention with 2 repetitions or 8 is determined by a drawing by lot after joint measurement has been done. Therapists who will oversee treatment and instruction first learn whether the group should be instructed in 2 or 8 repetitions at the first group training. The same applies to the included patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Range of Motion in knee joint | Day 1(baseline) and day 18
  Active flexion and extension measured with goniometer by physiotherapist (normal Range of motion (normal 0-140 degrees)

SECONDARY OUTCOMES:
6 minutes walk test | Day 1(baseline) and day 18
  How many meters can be walked in 6 minutes
30 seconds stand and sit test | Day 1(baseline) and day 18
  How many times can the person stand up and sit down without using hands
Numerical Rating Scale (NRS) | Day 1(baseline) and day 18
  Patients rating their pain from 0-10 on a scale (0=no pain/10=worst pain possible). Patients rates before - and after 6 minuts walking test
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | Day 1(baseline) and day 18
  Self-reported outcome measure assessing the patient's opinion about the health symptoms, and functionality of their knee (0-100 points - the higher score the better functionality)

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Mogensen, cand.scient., Study Director — Quality coordinator
Locations (1):
- Nordsjællands Hospital, Montebello, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beswick AD, Wylde V, Gooberman-Hill R, Blom A, Dieppe P. What proportion of patients report long-term pain after total hip or knee replacement for osteoarthritis? A systematic review of prospective studies in unselected patients. BMJ Open. 2012 Feb 22;2(1):e000435. doi: 10.1136/bmjopen-2011-000435. Print 2012. PMID 22357571
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Silva M, Shepherd EF, Jackson WO, Pratt JA, McClung CD, Schmalzried TP. Knee strength after total knee arthroplasty. J Arthroplasty. 2003 Aug;18(5):605-11. doi: 10.1016/s0883-5403(03)00191-8. PMID 12934213
- [Background] Gonzalez Della Valle A, Leali A, Haas S. Etiology and surgical interventions for stiff total knee replacements. HSS J. 2007 Sep;3(2):182-9. doi: 10.1007/s11420-007-9053-4. PMID 18751792
- [Background] Mutsuzaki H, Takeuchi R, Mataki Y, Wadano Y. Target range of motion for rehabilitation after total knee arthroplasty. J Rural Med. 2017 May;12(1):33-37. doi: 10.2185/jrm.2923. Epub 2017 May 24. PMID 28593015
- [Background] Matsuda S, Kawahara S, Okazaki K, Tashiro Y, Iwamoto Y. Postoperative alignment and ROM affect patient satisfaction after TKA. Clin Orthop Relat Res. 2013 Jan;471(1):127-33. doi: 10.1007/s11999-012-2533-y. PMID 22903282
- [Background] Maloney WJ. The stiff total knee arthroplasty: evaluation and management. J Arthroplasty. 2002 Jun;17(4 Suppl 1):71-3. doi: 10.1054/arth.2002.32450. PMID 12068410
- [Background] da Silva RR, Santos AA, de Sampaio Carvalho Junior J, Matos MA. Quality of life after total knee arthroplasty: systematic review. Rev Bras Ortop. 2014 Sep 19;49(5):520-7. doi: 10.1016/j.rboe.2014.09.007. eCollection 2014 Sep-Oct. PMID 26229855
- [Background] Liao CD, Tsauo JY, Huang SW, Chen HC, Chiu YS, Liou TH. Preoperative range of motion and applications of continuous passive motion predict outcomes after knee arthroplasty in patients with arthritis. Knee Surg Sports Traumatol Arthrosc. 2019 Apr;27(4):1259-1269. doi: 10.1007/s00167-018-5257-z. Epub 2018 Dec 7. PMID 30523369
- [Background] Sanchez Mayo B, Rodriguez-Mansilla J, Gonzalez Sanchez B. [Recovery from total knee arthroplasty through continuous passive motion]. An Sist Sanit Navar. 2015 May-Aug;38(2):297-310. doi: 10.23938/ASSN.0079. Spanish. PMID 26486536
- [Background] Joshi RN, White PB, Murray-Weir M, Alexiades MM, Sculco TP, Ranawat AS. Prospective Randomized Trial of the Efficacy of Continuous Passive Motion Post Total Knee Arthroplasty: Experience of the Hospital for Special Surgery. J Arthroplasty. 2015 Dec;30(12):2364-9. doi: 10.1016/j.arth.2015.06.006. Epub 2015 Jun 14. PMID 26165955
- [Background] Herbold JA, Bonistall K, Blackburn M, Agolli J, Gaston S, Gross C, Kuta A, Babyar S. Randomized controlled trial of the effectiveness of continuous passive motion after total knee replacement. Arch Phys Med Rehabil. 2014 Jul;95(7):1240-5. doi: 10.1016/j.apmr.2014.03.012. Epub 2014 Mar 28. PMID 24685389
- [Background] Harvey LA, Brosseau L, Herbert RD. Continuous passive motion following total knee arthroplasty in people with arthritis. Cochrane Database Syst Rev. 2014 Feb 6;2014(2):CD004260. doi: 10.1002/14651858.CD004260.pub3. PMID 24500904
- [Background] Boese CK, Weis M, Phillips T, Lawton-Peters S, Gallo T, Centeno L. The efficacy of continuous passive motion after total knee arthroplasty: a comparison of three protocols. J Arthroplasty. 2014 Jun;29(6):1158-62. doi: 10.1016/j.arth.2013.12.005. Epub 2013 Dec 14. PMID 24412145
- [Background] Trzeciak T, Richter M, Ruszkowski K. [Effectiveness of continuous passive motion after total knee replacement]. Chir Narzadow Ruchu Ortop Pol. 2011 Nov-Dec;76(6):345-9. Polish. PMID 22708322
- [Background] Bhave A, Sodhi N, Anis HK, Ehiorobo JO, Mont MA. Static progressive stretch orthosis-consensus modality to treat knee stiffness-rationale and literature review. Ann Transl Med. 2019 Oct;7(Suppl 7):S256. doi: 10.21037/atm.2019.06.55. PMID 31728380
- [Background] Bade MJ, Stevens-Lapsley JE. Early high-intensity rehabilitation following total knee arthroplasty improves outcomes. J Orthop Sports Phys Ther. 2011 Dec;41(12):932-41. doi: 10.2519/jospt.2011.3734. Epub 2011 Sep 30. PMID 21979411
- [Background] Mau-Moeller A, Behrens M, Finze S, Bruhn S, Bader R, Mittelmeier W. The effect of continuous passive motion and sling exercise training on clinical and functional outcomes following total knee arthroplasty: a randomized active-controlled clinical study. Health Qual Life Outcomes. 2014 May 9;12:68. doi: 10.1186/1477-7525-12-68. PMID 24886619
- [Background] Papotto BA, Mills T. Treatment of severe flexion deficits following total knee arthroplasty: a randomized clinical trial. Orthop Nurs. 2012 Jan-Feb;31(1):29-34. doi: 10.1097/NOR.0b013e3182419662. PMID 22278649
- [Background] Jakobsen TL, Christensen M, Christensen SS, Olsen M, Bandholm T. Reliability of knee joint range of motion and circumference measurements after total knee arthroplasty: does tester experience matter? Physiother Res Int. 2010 Sep;15(3):126-34. doi: 10.1002/pri.450. PMID 20024893
- See also: Danish knee arthroplasty register (2019) — http://docplayer.dk/161122569-Dansk-knaealloplastikregister.html
- See also: Organization for Danish physiotherapists - measuring tools — https://www.fysio.dk/fafo/maleredskaber/ledmaling-af-kna1